CLINICAL TRIAL: NCT07024576
Title: Preoperative Serial Casting, Stretching, and Massage Therapy Package for Dupuytren's Patients With Severe Proximal Interphalangeal Joint Contracture: A Feasibility Study Protocol for a Randomised Trial
Brief Title: Preoperative Serial Casting, Education, and Therapy for Dupuytren's Contracture
Acronym: PRESCET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Dorset County Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11151
Record Dates: First submitted 2025-05-27; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Dupuytren&Amp;#39;s Contracture; Dupuytren&Amp;#39;s Fasciectomy; Dupuytren&Amp;#39;s Disease
Keywords: Dupuytren's; Fasciectomy; Preoperative therapy

STUDY DESIGN:
Intervention Model Description: Two-arm randomised feasibility study
Who Masked: Outcomes Assessor
Masking Description: Surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A serial casting intervention protocol involving the application of heat, stretching, and massage before casting. This is repeated weekly for four weeks, with the cast removed and reapplied each time to promote gradual elongation of restricted tissue. Additionally, they will receive an education session covering disease pathology, surgical objectives, postoperative expectations, pain, and recovery milestones.
  Interventions: Other: Preoperative casting intervention
- Control group (No Intervention): An education session covering disease pathology, surgical objectives, postoperative expectations, pain, and recovery milestones only, with no added preoperative therapy.

INTERVENTIONS:
Other: Preoperative casting intervention — A serial casting intervention protocol involving the application of heat, stretching, and massage before casting. This is repeated weekly for four weeks, with the cast removed and reapplied each time to promote gradual elongation of restricted tissue.
  Arms: Intervention group

SUMMARY:
We are running a small study to test whether a special type of therapy - including casting, stretching, and massage - might help improve recovery after Dupuytren's Fasciectomy.

The study is taking place at Dorset County Hospital and will involve people who are already scheduled for surgery and have a permanent bend of 30 degrees or more in the middle joint of one or more fingers.

The therapy will be given before surgery to see if it helps people get a better result afterwards.

We want to find out:

* Who would be suitable to take part in a future, larger study
* Which results are most important to measure (like finger movement or grip strength)
* How many people complete the full therapy and follow-up We'll also speak to patients and healthcare professionals to understand how acceptable and practical this therapy is.

The goal is to see whether it's possible and worthwhile to run a larger study in the future, to find out if pre-surgery therapy can become a helpful part of treatment for people undergoing Dupuytren's Fasciectomy.

DETAILED DESCRIPTION:
Dupuytren's disease is a common and progressively disabling condition affecting the connective tissue of the palm of the hand. It causes fibrosis of the palmar fascia, which can lead to one or more fingers becoming incapable of full extension, adopting a fixed flexion contracture. This loss of extension can significantly impair hand function and limit daily activities. While surgery (typically fasciectomy) remains the most effective treatment for Dupuytren's contracture, outcomes are often less favourable when the deformity involves the proximal interphalangeal joint, particularly in severe cases where the contracture exceeds 30 degrees.

This feasibility study investigates whether a short course of preoperative therapy, delivered before surgery, can help improve recovery and outcomes after Dupuytren's Fasciectomy. The intervention includes:

* Heat application
* Stretching and massage
* Serial casting - a method of gently lengthening tight tissue by applying and adjusting a soft cast weekly prior to surgery The treatment is designed to gently lengthen tight tissues and increase joint range of movement in the affected fingers prior to surgery, with the goal of improving movement and function after surgery.

We are recruiting approximately 20 adult patients from Dorset County Hospital NHS Foundation Trust who:

* Are scheduled for Dupuytren's Fasciectomy
* Have a PIP joint contracture of 30 degrees or more

Participants will be randomly assigned to one of two groups:

* Intervention group: Will receive the four-week preoperative therapy programme plus an education session covering disease pathology, surgical objectives, postoperative expectations, pain, and recovery milestones.
* Control group: Will receive the same education programme only, with no added preoperative therapy.

After surgery, all participants will follow standard postoperative therapy and attend follow-up appointments up to 12 weeks post-op, where we will collect outcome measures including:

* Finger range of motion
* Hand function (using the Michigan Hand Outcomes Questionnaire - MHQ)
* Grip strength
* Patient satisfaction
* Completion and retention rates throughout the study To understand how practical and acceptable this approach is in real-world clinical settings, we will also conduct interviews with patients and healthcare professionals to explore their experiences and suggestions for improvement.

As a feasibility study, the goal is not to test effectiveness, but to assess whether a larger, definitive trial is achievable. Specifically, we aim to:

* Determine who is suitable and willing to take part
* Identify the most relevant outcome measures
* Evaluate participation and follow-up rates
* Understand acceptability from both patients and clinicians
* Estimate the resources and planning needed for a full-scale trial If this study shows that the intervention is feasible and well-received, we aim to proceed with a multi-centre randomised controlled trial to evaluate the effectiveness of preoperative therapy as part of standard care for Dupuytren's fasciectomy.

This research is a collaboration between Dorset County Hospital NHS Foundation Trust and Bournemouth University, with active involvement and guidance from a Patient and Public Involvement steering group made up of individuals with lived experience of Dupuytren's disease and the healthcare professionals involved in their care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or older.
* One or more fingers with a Dupuytren's flexion contracture greater than 30° at the PIP joint.
* Awaiting fasciectomy surgery for Dupuytren's contracture.
* Willing and able to provide informed consent for participation in the study.

Exclusion Criteria:

* Individuals awaiting needle fasciotomy, dermofasciectomy, or segmental fasciectomy.
* A history of previous treatment for Dupuytren's contracture (e.g., surgery, collagenase injection, or needle fasciectomy) to the study reference digit.
* A history of any other pre-existing hand disorder causing significant movement restriction, pain, or affecting hand function (e.g., post-traumatic stiffness, arthritis, infection).
* Non-English speaking participants due to the need for completing multiple questionnaires that have not been validated in multiple languages.
* Inability to attend follow-up appointments within the required timeframes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression criteria assessment | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Primary Outcome Measure:
  Feasibility of progressing to a full randomised controlled trial (RCT) based on predefined progression criteria across eight domains. These include participant availability (≥37 listed for fasciectomy over 9 months), eligibility rate (≥54%), consent rate among eligible participants (≥80%), and willingness to undergo randomisation (≥80%). Additional feasibility indicators include the ability to maintain blinding of assessors and surgeons throughout the study, high intervention acceptability determined via qualitative evaluation, adherence to preoperative splinting (>80%), and retention at 12-week follow-up (>80%). Safety is assessed by tracking adverse events, with progression supported if ≤20% of participants experience an adverse reaction. Thresholds for "Go," "Amend," or "Stop" decisions are defined for each domain.

SECONDARY OUTCOMES:
Active range of movement of the affected finger(s) | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Active range of movement of the affected finger(s), recorded individually at the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints. Measurements are obtained using a standard manual goniometer, with the participant seated, forearm supported in neutral rotation, and wrist in a neutral position.
  * Flexion is defined as the angle at each joint when the participant actively attempts to flex the finger (i.e., make a fist), measured from the neutral (0°) position toward full flexion.
  * Extension is defined as the angle achieved at each joint when the participant actively attempts to fully straighten the finger, measured from the neutral position toward full extension or hyperextension.
  Each joint is measured and recorded separately in degrees for both maximal flexion and maximal extension. AROM is assessed at baseline, at each preoperative visit, and at 12 weeks postoperatively.
Passive range of movement (PROM) of the affected finger(s) | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Passive range of movement (PROM) of the affected finger(s), recorded individually at the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints. Measurements are obtained using a standard manual goniometer, with the participant seated, forearm supported in neutral rotation, and wrist in a neutral position.
  * Passive flexion is defined as the angle at each joint achieved when the examiner passively moves the finger into maximal flexion without patient effort, measured from the neutral (0°) position.
  * Passive extension is defined as the angle at each joint when the examiner passively moves the finger into full extension or hyperextension, again without patient effort.
  Each joint is measured and recorded separately in degrees for both maximal passive flexion and maximal passive extension. PROM is assessed at baseline, at each preoperative visit, and at 12 weeks postoperatively.
Grip strength of the affected hand | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Grip strength of the affected hand is measured using a Jamar hydraulic hand dynamometer. Strength is assessed in kilograms (kg) with the participant seated, shoulder adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral position, and wrist positioned between 0-30° extension and 0-15° ulnar deviation.
  Participants are instructed to squeeze the dynamometer maximally for 3 seconds. Three trials are performed with a 30-second rest between attempts, and the mean value of the three trials is recorded. The second handle position on the Jamar dynamometer is used for consistency.
  Grip strength is measured at baseline, at each preoperative visit, and at 12 weeks postoperatively. Measurements at baseline and 12 weeks postoperatively are performed by therapists blinded to group allocation, using standardised equipment and procedures to ensure reliability and comparability across time points.
Michigan Hand Questionnaire (MHQ) | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Hand function is assessed using the Michigan Hand Questionnaire (MHQ), a validated, condition-specific, patient-reported outcome measure. The MHQ evaluates six domains: hand function, activities of daily living (ADLs), pain, work performance, aesthetics, and satisfaction with hand function. It consists of 37 items, each domain scored on a 0 to 100 scale. For all domains except pain, higher scores indicate better outcomes; in the pain domain, higher scores reflect greater pain.
  Participants complete the MHQ at baseline, at each preoperative visit, and at 12 weeks postoperatively. The questionnaire is administered by a therapist, who reads each question aloud and records the participant's responses directly onto the form, following the standardised MHQ scoring protocol.
Patient-Specific Functional Scale (PSFS) | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Hand function is also assessed using the Patient-Specific Functional Scale (PSFS). The PSFS is a validated, patient-reported outcome measure used to evaluate functional limitations specific to the individual's condition. Participants are asked to identify up to three activities that they are currently unable to perform or perform with difficulty due to their hand condition.
  Each activity is rated on a 0 to 10 numeric rating scale, where 0 represents "unable to perform the activity" and 10 represents "able to perform the activity without any difficulty." Scores are recorded for each activity, and an average score is calculated to reflect overall functional ability.
  The PSFS is administered at baseline, at each preoperative visit, and at 12 weeks postoperatively. This outcome measure captures patient-defined functional goals and changes over time, providing a highly individualised and responsive assessment of functional improvement
Barriers and facilitators to adherence | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  Barriers and facilitators to attainment of the intervention, identified through semi-structured qualitative interviews with both participants and healthcare professionals involved in the trial. Interviews are conducted to explore individual and system-level factors that influence engagement with and delivery of the intervention, including adherence, acceptability, perceived benefit, and contextual constraints.
  Interviews are conducted at the end of the intervention period with a selection of participants using a topic guide developed from existing literature and trial objectives, and are audio-recorded, transcribed verbatim, and anonymised. Data are analysed thematically using framework analysis to identify recurring themes related to barriers and facilitators to intervention delivery and uptake.
Sample size estimation | From enrolment 4 weeks preoperatively, till final follow-up at 12 weeks postoperatively
  The sample size estimation for a future definitive trial will be informed by the distribution and completeness of outcome data, and by recruitment, consent, adherence, and retention rates observed during the trial. These estimates will be used to model various trial design scenarios, ensuring adequate power to detect clinically meaningful differences in a future randomised controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Crook, Principal Investigator — Dorchester County Hospital
Locations (1):
- Dorchester County Hospital NHS Foundation Trust, Dorchester, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The findings of the trial will be made publicly available through publication or other dissemination tools without any unnecessary delay. Datasets will be made available by the corresponding author on reasonable request and in accordance with consent and ethical approval.

REFERENCES:
- [Background] Mellor K, Albury C, Dutton SJ, Eldridge S, Hopewell S. Recommendations for progression criteria during external randomised pilot trial design, conduct, analysis and reporting. Pilot Feasibility Stud. 2023 Apr 15;9(1):59. doi: 10.1186/s40814-023-01291-5. PMID 37061720